CLINICAL TRIAL: NCT06358300
Title: Visceral Adiposity Index Levels in Polycystic Ovary Syndrome Subtypes
Brief Title: Visceral Adiposity Index Differences Between Subtypes of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Sponsor
Other Study IDs: Usakpcos2
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Visceral Adiposity Index; Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Visceral Adiposity Index; PCOS Subtypes
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples Without DNA — After 8-12 hours of fasting, 2-3 ml of blood will be taken for serum HDL and TG measurement. Blood will be centrifuged and frozen at -70 °C.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Controls: Healthy controls between aged 18-35 years
- PCOS Subtype 1: Hyperandrogenemia+oligoanovulation+PCO appearance on USG
- PCOS Subtype 2: Hyperandrogenemia+oligoanovulation
- PCOS Subtype 3: Hyperandrogenemia+PCO appearance on USG
- PCOS Subtype 4: Oligoanovulation+PCO appearance on USG

SUMMARY:
We aimed to investigate visceral adiposity index (VAI) in patients with different phenotype of policystic ovary syndrome (PCOS) and to compare healthy controls.

DETAILED DESCRIPTION:
Polycystic ovary syndrome; Metabolic disorders such as insulin resistance, dyslipidemia, glucose intolerance, hypertension and obesity are often accompanied, and increased inflammation is the main characteristic of this syndrome. While the presence or absence of PCOS was important until recently, recent studies have shown that metabolic changes and inflammation occur at different degrees in different subtypes of PCOS. Therefore, PCOS cases are divided into 4 subtypes. These; Subtype 1 has hyperandrogenemia + oligoanovulation + PCO appearance on ultrasonography (USG), Subtype 2 has hyperandrogenemia + oligoanovulation, Subtype 3 has hyperandrogenemia + PCO appearance on USG, and Subtype 4 has oligoanovulation + PCO appearance on USG. As the subtype number of polycystic ovary syndrome decreases, the severity and frequency of metabolic disorders and inflammation accompanying polycystic ovary syndrome increase.

Patients with polycystic ovary syndrome often have abdominal obesity, which leads to hypertension, dyslipidemia, impaired glucose tolerance, Type 2 Diabetes and metabolic syndrome, which predisposes to the development of cardiovascular disease. Visceral adiposity is associated with abnormal lipid levels, proinflammatory activity, insulin resistance, and hyperandrogenism. Increased visceral adiposity increases the risk of metabolic syndrome, Type 2 Diabetes, and cardiovascular events in women with PCOS; It also aggravates ovulation dysfunction and hyperandrogenism.

Visceral adiposity index (VAI) is a simple marker of visceral adipose tissue dysfunction and visceral adiposity and is associated with insulin resistance, hyperinsulinemia, hyperandrogenism and anovulation. Visceral adiposity index (VAI) is one of the new methods used to determine visceral adiposity and predict cardiometabolic risks in patients. Visceral adiposity index is the strongest marker determining metabolic syndrome in both obese and non-obese PCOS patients. Visceral adiposity index is calculated with the formula [Waist circumference / (36.58 + (1.88xBMI)] x (Triglyceride/0.81) x (1.52/HDL-C). Visceral adiposity index is used in the clinical presentations of PCOS and treatment success. It is reported to be a useful marker that enables early detection and intervention of the risk of metabolic syndrome in women. Since there are different metabolic effects in different subtypes of PCOS, we aimed to investigate whether there is a difference between visceral adiposity indexes in different PCOS subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who applied for reasons such as hair growth, acne, menstrual irregularity or infertility and were diagnosed with PCOS after examination, biochemical, hormonal and sonographic tests,
2. Female patients between the ages of 18-35,
3. Patients without known cancer, liver or kidney failure,
4. Patients who do not take medications that will affect HDL, TG levels and insulin resistance,
5. Female patients without active infection will be included. -

Exclusion Criteria:

1. Female patients under eighteen years of age and >35 years of age,
2. Patients with known cancer, liver and kidney failure,
3. Patients taking medications that will affect HDL, TG levels and insulin resistance,
4. Patients with active infection will not be included in the study. -

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Woman aged between 18 and 35, age-matched between groups, diagnosed with PCOS and without a known cancer diagnosis, liver and kidney failure, not taking medications that would affect HDL, TG levels and insulin resistance and without active infection.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Visceral Adiposity Index Differences Between Subtypes of Polycystic Ovary Syndrome | Eight months
  Since there are different metabolic effects in different subtypes of polycystic ovary syndrome; In this study we aimed to investigate whether there is a difference between VAI in different PCOS subtypes and the difference between these subtypes and the healthy group.

CONTACTS AND LOCATIONS:
Locations (1):
- Usak Training and Research Hospital, Uşak, Turkey (Türkiye)